CLINICAL TRIAL: NCT03346551
Title: Postnatal Depression, Attachment and Self-defining Memories
Acronym: PNDattachMEMO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PA17012
Record Dates: First submitted 2017-10-23; First posted 2017-11-17 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Postnatal Depression
Keywords: Postnatal depression; Attachment; Self-defining memories
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- women with postnatal depression (Experimental)
  Interventions: Behavioral: Evaluation of the quality attachment : "Adult Attachment Narratives" and "CaMir scale"; Behavioral: Evaluation of the self-defining memories : "Specific Questionnaire during an interview"
- women without postnatal depression (Other)
  Interventions: Behavioral: Evaluation of the quality attachment : "Adult Attachment Narratives" and "CaMir scale"; Behavioral: Evaluation of the self-defining memories : "Specific Questionnaire during an interview"

INTERVENTIONS:
Behavioral: Evaluation of the quality attachment : "Adult Attachment Narratives" and "CaMir scale" — Evaluation of the quality attachment : "Adult Attachment Narratives" and "CaMir scale"
Behavioral: Evaluation of the self-defining memories : "Specific Questionnaire during an interview" — Evaluation of the self-defining memories : "Specific Questionnaire during an interview"

SUMMARY:
The specificity of postnatal depression (PND) was acted as full entity within the depressions, by B. Pitt in 1968, through the description of a specific nosography which describes "an atypical depression of the post-partum ".

Actually, the epidemiological studies agree on prevalence from 10 to 15 % of PND. With two peaks of frequency, the first one around the 6th and 12th week comment native and the second during the second half-year. This rate of PND represents in France 75000 to 100000 women a year.

The professionals of the perinatal period are interested in this disorder because of the consequences for the woman herself, and of the impact on the premature interactions mother-baby. These interactions and the direct effects of the PND on the mother will have for influence an important slowing down on the development of the baby. Moreover, the study of Lemaitre and Candilis in 1999, brings the figure of 15 % of the PND which will have an impact on the development of the baby.

The sensation of the depression testifies of a process of change and of psychic conflict favored by the psychic transparency of the pregnancy.

Although the first treaty on this specific nosography dates more than 150 years of numerous questions stay suspends it.

These questions and the reflections which surround them found on their path tools ensuing from the theory of the attachment, formalized by John Bowlby. For more than three decades, these profiles of attachment, specified by Mary Ainsworth: secure, anxious-ambivalent, anxious-avoided and disorganized later, disrupted, is studied, estimated and their evolution during a life is observed. Thanks to these models well known for the same person at a time t, it is now their effects in the interpersonal relations which are studied. Between the people but also on the person himself, its image of her, and its autobiographical memory.

The autobiographical memory represents a central component of the human memory. At a very general level, it's possible to define it as the capacity of a person to remember its past experiences. The review of the literature on the functioning of the episodic autobiographical memory during the depression highlights three main results: the too bi generalization of the memories, the congruence in the humor and the frequency of the intrusive memories characterized by an involuntary reminder, fast and effortlessly (Lemogne and al., 2006; Lemogne and al., 2012). The authors specify that there are links between strategies of avoidance of the intrusive memories and the phenomenon of generalization. These links ask to be explored within a model integrating, self and episodic autobiographical memory in the field of the depression. The use of the memories defining the one could allow to study more specifically this kind of memories. The memories defining the one were introduced to Ape and Moffitt (1991) to characterize a specific category of autobiographical memories. The memories defining the one are important personal memories which help a person to understand whom this person is as individual. In a way, they build the life story and support the personal identity. Connected to other similar memories, the self-defining memories contain numerous sensory details and are often associated to a strong emotional charge. They are also connected to long-term purposes, to concerns or to unsolved conflicts.

Recent studies used the self-defining memories (French version adapted by Mr van der Linden's team, Switzerland) as tool to understand better the psychological disorders from which certain people suffer. The studies show that the self-defining memories undergo modifications the characteristics of which are in connection with every pathology (works of the team of J.M. Danion).

In 1994, Moffit and al. studied a group of students with evaluation of the depressive symptomatology. They established that the presenting subjects of high scores of depression develop more generalized memories than the other participants when is asked to them a self-defining memorie positive. For the memories with negative valence, no difference is found among the tested students. There are no data in the literature on the self-defining memories and the postnatal depression. Besides, there is only a single search, not published which explores the links between the attachment and the memories defining the one (Tagini, Conway and Meins, looks for not published, quoted by Conway, to Ape and Tagini, on 2004). The authors present the results according to the styles of attachment. So, autobiographical memories would vary according to the cognitive and emotional dimensions, in connection with differences in the style of attachment. In every style of attachment would correspond certain specificities in the contents and in the form of the self-defining memories.

DETAILED DESCRIPTION:
In this context, it seems important to look for if there are specificities concerning the profiles of attachment and the self-defining memories at the patients suffering from postnatal depression. Especially as the current literature approaches only little this subject of public health.

To analyze these specificities, two groups (group postnatal depression versus group control) will compare by estimating the type of maternal attachment and theirs self-definig memories, without omitting to look for a possible psychiatric pathology, and a personality problem at the mother.

The main objective of this study will be to highlight specificities of the style of attachment and the personal identity in the postnatal depression.

The secondary objectives of this study will on one hand be to look for the existence of links between the various clinical variables in the postnatal depression.

And on the other hand to look for psychological and clinical factors which can be markers of vulnerability and\or factors of protection of the depression comment native (comparison between both groups of subjects).

The participation to this study will be proposed to all the women of both centers, throughout the inclusion. Those who will have accepted will fill a scale Edinburgh Post-natal Depression Scale (EPDS). The score which will decide in which group women will be assigned :

* < 11 group control
* > 11 group PND The specific visit in the study will take place in a identical way for the cases and the witnesses.

The patients will be seen at first by a doctor a child psychiatrist who will make a data collection sociodemographic and clinical and the signing of various questionnaires : Mini International Neurospychiatric Interview (MINI), Adult Attachment Narratives (AAN), Camir scale and Perceived Social Support Questionnaire (QSSP).

Secondly, the patients will be seen by a psychologist to pursue the clinical evaluation (Trait Anxiety Inventory (STAI), Beck Depression Inventory and self-esteem scale (EES), Scale of vocabulary (MILL-HILL) and to realize the signing of the questionnaire of the self-defining memories.

ELIGIBILITY:
inclusion criteria :

* Group 1 : women with postnatal depression
* Group 2 : women without postnatal depression
* women consenting to participate to the study
* women enrolled in the national healthcare insurance program
* women older than 18 years old

exclusion criteria :

* women younger than 18 years old
* women protected by the law

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-10-13 (Actual); Primary Completion 2019-11-13 (Estimated); Study Completion 2019-12-13 (Estimated)

PRIMARY OUTCOMES:
Quality attachment | Day 0
  Evaluation of the quality attachment using "Adult Attachment Narratives"
Quality attachment | Day 0
  Evaluation of the quality attachment using "CaMir scale"

SECONDARY OUTCOMES:
First Self-defining memory | Day 0
  Evaluation of the self-defining memory using a specific questionnaire from Singer, J. A., & Moffitt, K. H. (1991-1992) and Thorne, A., & McLean, K. C. (2001), translate in French
Second Self-defining memory | Day 0
  Evaluation of the self-defining memory using a specific questionnaire from Singer, J. A., & Moffitt, K. H. (1991-1992) and Thorne, A., & McLean, K. C. (2001), translate in French
Third Self-defining memory | Day 0
  Evaluation of the self-defining memory using a specific questionnaire from Singer, J. A., & Moffitt, K. H. (1991-1992) and Thorne, A., & McLean, K. C. (2001), translate in French

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France

IPD SHARING:
Plan to Share IPD: No